CLINICAL TRIAL: NCT03081403
Title: Quantitative Sensory Testing in Subjects With Sensitive Skin or Not
Acronym: SENSISKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SENSISKIN 29CRB16.0100
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Sensitive Skin
Keywords: Sensitive skin; Quantitative Sensory Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with sensitive skin (Other): Subjects with a score greater than 50 on the sensitive scale
  Interventions: Device: Quantitative Sensory Testing
- Subjects without sensitive skin (Other): Subjects with result lower than 20 on the sensitive scale
  Interventions: Device: Quantitative Sensory Testing

INTERVENTIONS:
Device: Quantitative Sensory Testing — Study of detection thresholds of vibration, cold and pain related to the heat in the dominant hand of the subjects through the QST.

SUMMARY:
Sensitive skin is a common problem, with 50% of women and 30% of men in Europe feel they have sensitive skin.

The Quantitative sensory testing (QST) is a physico-psychic method that uses gradients stimuli of different modalities to measure a subjective somatosensory response. This allows to characterize sensory dysfunction by assessing the participation of small and large nerve fibers.

The aim of this project is to characterize the presence or absence of a neurological disorder in patients with sensitive skin. This discovery would be a decisive argument to reinforce the suspicion that sensitive skins is linked to a small fiber neuropathy.

DETAILED DESCRIPTION:
Sensitive skin is a common problem, with 50% of women and 30% of men in Europe feel they have sensitive skin. A sensitive skin is characterized by the occurrence of tingling sensations, tightness, heat, burning, itching or pain triggered by non pathogenic factors such as wind, heat, cold, water , cosmetics, toiletries, stress...

The Quantitative sensory testing (QST) is a physico-psychic method that uses gradients stimuli of different modalities to measure a subjective somatosensory response. This allows to characterize sensory dysfunction by assessing the participation of small and large nerve fibers.

The aim of this project is to characterize the presence or absence of a neurological disorder in patients with sensitive skin. This discovery would be a decisive argument to reinforce the suspicion that sensitive skins is linked to a small fiber neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 20 and 60 years
* Cooperating patient
* Informed and written consent of the subject
* Affiliated to the social security
* For subjects with sensitive skin:

subjects with a score greater than 50 on the scale sensitive scale

- To control subjects: subjects with result of less than 20 sensitive to the scale scale

Exclusion Criteria:

* Adults subject with legal protection
* Subject in a social institution.
* Subject with major cognitive or psychiatric disorders
* Subject with pathological use of alcohol or consumption of another drug.
* Subject with skin involvement of the back of the dominant hand or malformation.
* Known sensitive neuropathy
* Pregnant woman
* Subject receiving medical treatment which may interfere with the results.
* Subject with treatment in the back of the dominant hand.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Cutaneous perception threshold | 6 months
  The cutaneous perception threshold of pain to heat.

SECONDARY OUTCOMES:
The cutaneous perception threshold of vibration | 6 months
  The cutaneous perception threshold of pain to harm.
The cutaneous perception threshold of cold | 6 months
  The cutaneous perception threshold of cold

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No